CLINICAL TRIAL: NCT01131260
Title: A Randomized Trial of Fetal ECG ST Segment and T Wave Analysis as an Adjunct to Electronic Fetal Heart Rate Monitoring (STAN)
Brief Title: Fetal ST Segment and T Wave Analysis in Labor
Acronym: STAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The George Washington University Biostatistics Center (Other)
Collaborators: Neoventa Medical (Unknown); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HD36801-STAN; U10HD021410 (NIH); U10HD027869 (NIH); U10HD027917 (NIH); U10HD053118 (NIH); U10HD027915 (NIH); U10HD034208 (NIH); U10HD053097 (NIH); U10HD040500 (NIH); U10HD040485 (NIH); U10HD040544 (NIH); U10HD040545 (NIH); U10HD040560 (NIH); U10HD040512 (NIH); U01HD036801 (NIH); U10HD068268 (NIH); U10HD068282 (NIH)
Record Dates: First submitted 2010-05-25; First posted 2010-05-26 (Estimated); Results first posted 2019-04-05 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Pregnancy; Obstetric Labor; Parturition
Keywords: STAN; Fetal monitoring; Fetal acidosis; Fetal heart rate monitoring; Perinatology

STUDY DESIGN:
Intervention Model Description: The study is a randomized, controlled clinical trial of 11,000 women in labor at > 36.0 weeks gestation randomized to one of two groups using the STAN S31 system:
  * Fetal STAN electrode inserted and data available to caregivers (open device group)
  * Fetal STAN electrode inserted, but data masked to the caregivers (masked device group)
Who Masked: Care Provider
Masking Description: The study is a randomized, controlled clinical trial of 11,000 women in labor at > 36.0 weeks gestation randomized to one of two groups using the STAN S31 system:
  * Fetal STAN electrode inserted and data available to caregivers (open device group)
  * Fetal STAN electrode inserted, but data masked to the caregivers (masked device group)
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Open Group (Experimental): • Fetal STAN monitor electrode inserted and data available to caregivers
  Interventions: Device: fetal STAN monitor
- Masked Group (Other): •Fetal STAN monitor electrode inserted, but data masked to the caregivers
  Interventions: Device: fetal STAN monitor

INTERVENTIONS:
Device: fetal STAN monitor — The STAN monitor is a system for fetal surveillance that displays the FHR, the uterine activity and information resulting from the analysis of the ST segment of the fetal ECG.
  Other Names: STAN S31

SUMMARY:
The purpose of this research is to test a new instrument, called a fetal STAN monitor, that may be used during labor to monitor the electrical activity of the baby's heart. This new instrument is designed to help the doctor determine how well the baby is doing during labor. It will be used along with the existing electronic fetal monitor used to measure the baby's heart rate and the mother's contractions during birth. The specific purpose of this research study is to see if this new instrument (fetal STAN monitor) will have an impact on newborn health.

DETAILED DESCRIPTION:
A Randomized Trial of Fetal ECG ST Segment and T Wave Analysis as an Adjunct to Electronic Fetal Heart Rate Monitoring (STAN):

Fetal ECG analysis of the ST segment (STAN) is now FDA-approved and clinically available in the United States as an adjunct for the interpretation of electronic fetal heart rate patterns. There have been a number of randomized controlled trials as well as observational studies in Europe documenting utility of this modality in terms of reducing fetal acidosis at birth, and decreasing the need for operative vaginal delivery. However, despite these endorsements, there remain concerns with the application of the technology to the United States. None of the randomized trials were performed in the United States where patient case-mix and obstetrical practice, such as the use of fetal scalp pH, differ from Europe, which may affect the impact of this technology on perinatal outcomes. Moreover, the results of the European studies are not uniformly positive.

This protocol describes a randomized controlled trial of the STAN technology as an adjunct to electronic fetal heart rate monitoring versus fetal heart rate monitoring alone.

ELIGIBILITY:
Inclusion Criteria:

* Singleton, cephalic pregnancy
* Gestational age at least 36 weeks, 1 day
* Cervical dilation of at least 2 cm and no more than 7 cm
* Ruptured membranes

Exclusion Criteria:

* Multifetal gestation
* Planned cesarean delivery
* Need for immediate delivery
* Absent variability or sinusoidal pattern at any time, or a Category II fetal heart rate pattern with absent variability in the last 20 minutes before randomization
* Inability to obtain or maintain an adequate signal within 3 trials of electrode placements
* Occurrence of any ST event during attempt to obtain adequate signal
* Patient pushing in the first stage of labor
* Known major fetal anomaly or fetal demise
* Previous uterine surgery
* Placenta previa on admission
* Maternal fever greater than or equal to 38 C or 100.4 F
* Active HSV infection
* Known HIV or hepatitis infection
* Other maternal and fetal contraindications for using the STAN monitor
* Enrollment in another labor study
* Participation in this trial in a previous pregnancy
* No certified or authorized provider available

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 11108 (Actual)
Dates: Start 2010-11; Primary Completion 2014-04 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Menachem Miodovnik, MD, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD); Rebecca Clifton, PhD, Principal Investigator — George Washington University Biostatistics Center; George Saade, MD, Study Chair — University of Texas; Michael Belfort, MD, Study Chair — University of Utah
Locations (13):
- United States (13):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Northwestern University, Chicago, Illinois
  - Wayne State University - Hutzel Hospital, Detroit, Michigan
  - Columbia University, New York, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Case Western University, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pittsburgh - Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Brown University, Providence, Rhode Island
  - University of Texas - Galveston, Galveston, Texas
  - University of Texas - Houston, Houston, Texas
  - University of Utah Medical Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
The dataset will be shared per NIH policy after the completion and publication of the main analyses. Requests for datasets can be sent to mfmudatasets@bsc.gwu.edu

REFERENCES:
- [Background] Rosen KG, Kjellmer I. Changes in the fetal heart rate and ECG during hypoxia. Acta Physiol Scand. 1975 Jan;93(1):59-66. doi: 10.1111/j.1748-1716.1975.tb05790.x. PMID 1155132
- [Background] Rosen KG, Isaksson O. Alterations in the fetal heart rate and ECG correlated to glycogen, creatine phosphate and ATP levels during graded hypoxia. Biol Neonate 1976;30:17-24
- [Background] Hokegard KH, Eriksson BO, Kjellmer I, Magno R, Rosen KG. Myocardial metabolism in relation to electrocardiographic changes and cardiac function during graded hypoxia in the fetal lamb. Acta Physiol Scand. 1981 Sep;113(1):1-7. doi: 10.1111/j.1748-1716.1981.tb06853.x. PMID 7315431
- [Background] Hokegard KH, Karlsson K, Kjellmer I, Rosen KG. ECG-changes in the fetal lamb during asphyxia in relation to beta-adrenoceptor stimulation and blockade. Acta Physiol Scand. 1979 Feb;105(2):195-203. doi: 10.1111/j.1748-1716.1979.tb06331.x. PMID 33536
- [Background] Dagbjartsson A, Herbertsson G, Stefansson TS, Kjeld M, Lagercrantz H, Rosen KG. Beta-adrenoceptor agonists and hypoxia in sheep fetuses. Acta Physiol Scand. 1989 Oct;137(2):291-9. doi: 10.1111/j.1748-1716.1989.tb08750.x. PMID 2618763
- [Background] Widmark C, Jansson T, Lindecrantz K, Rosen KG. ECG waveform, short term heart rate variability and plasma catecholamine concentrations in response to hypoxia in intrauterine growth retarded guinea-pig fetuses. J Dev Physiol. 1991 Mar;15(3):161-8. PMID 1940143
- [Background] Greene KR, Dawes GS, Lilja H, Rosen KG. Changes in the ST waveform of the fetal lamb electrocardiogram with hypoxemia. Am J Obstet Gynecol. 1982 Dec 15;144(8):950-8. doi: 10.1016/0002-9378(82)90190-9. PMID 7148927
- [Background] Rosen KG, Dagbjartsson A, Henriksson BA, Lagercrantz H, Kjellmer I. The relationship between circulating catecholamines and ST waveform in the fetal lamb electrocardiogram during hypoxia. Am J Obstet Gynecol. 1984 May 15;149(2):190-5. doi: 10.1016/0002-9378(84)90197-2. PMID 6720798
- [Background] Greene KR, Rosen KG. Long-term ST waveform changes in the ovine fetal electrocardiogram: the relationship to spontaneous labour and intrauterine death. Clin Phys Physiol Meas. 1989;10 Suppl B:33-40. doi: 10.1088/0143-0815/10/4b/005. PMID 2630159
- [Background] Widmark C, Hokegard KH, Lagercrantz H, Lilja H, Rosen KG. Electrocardiographic waveform changes and catecholamine responses during acute hypoxia in the immature and mature fetal lamb. Am J Obstet Gynecol. 1989 May;160(5 Pt 1):1245-50. doi: 10.1016/0002-9378(89)90204-4. PMID 2729402
- [Background] Gelli MG, Bergstrom J, Hultman E, Thalme B. Heart muscle and plasma electrolytes in normal and glucose-loaded rabbit foetuses under anoxia. Acta Obstet Gynecol Scand. 1969;48(1):34-55. doi: 10.3109/00016346909156625. No abstract available. PMID 5372122
- [Background] Rosen KG, Hokegard KH, Kjellmer I. A study of the relationship between the electrocardiogram and hemodynamics in the fetal lamb during asphyxia. Acta Physiol Scand. 1976 Nov;98(3):275-84. doi: 10.1111/j.1748-1716.1976.tb10312.x. PMID 11642
- [Background] Watanabe T, Okamura K, Tanigawara S, Shintaku Y, Akagi K, Endo H, Yajima A. Change in electrocardiogram T-wave amplitude during umbilical cord compression is predictive of fetal condition in sheep. Am J Obstet Gynecol. 1992 Jan;166(1 Pt 1):246-55. doi: 10.1016/0002-9378(92)91867-a. PMID 1733202
- [Background] Westgate JA, Bennet L, Brabyn C, Williams CE, Gunn AJ. ST waveform changes during repeated umbilical cord occlusions in near-term fetal sheep. Am J Obstet Gynecol. 2001 Mar;184(4):743-51. doi: 10.1067/mob.2001.111932. PMID 11262482
- [Background] Westgate J, Harris M, Curnow JS, Greene KR. Plymouth randomized trial of cardiotocogram only versus ST waveform plus cardiotocogram for intrapartum monitoring in 2400 cases. Am J Obstet Gynecol. 1993 Nov;169(5):1151-60. doi: 10.1016/0002-9378(93)90273-l. PMID 8238177
- [Background] Amer-Wahlin I, Hellsten C, Noren H, Hagberg H, Herbst A, Kjellmer I, Lilja H, Lindoff C, Mansson M, Martensson L, Olofsson P, Sundstrom A, Marsal K. Cardiotocography only versus cardiotocography plus ST analysis of fetal electrocardiogram for intrapartum fetal monitoring: a Swedish randomised controlled trial. Lancet. 2001 Aug 18;358(9281):534-8. doi: 10.1016/s0140-6736(01)05703-8. PMID 11520523
- [Background] Ojala K, Vaarasmaki M, Makikallio K, Valkama M, Tekay A. A comparison of intrapartum automated fetal electrocardiography and conventional cardiotocography--a randomised controlled study. BJOG. 2006 Apr;113(4):419-23. doi: 10.1111/j.1471-0528.2006.00886.x. PMID 16553653
- [Background] Vayssiere C, David E, Meyer N, Haberstich R, Sebahoun V, Roth E, Favre R, Nisand I, Langer B. A French randomized controlled trial of ST-segment analysis in a population with abnormal cardiotocograms during labor. Am J Obstet Gynecol. 2007 Sep;197(3):299.e1-6. doi: 10.1016/j.ajog.2007.07.007. PMID 17826428
- [Background] Noren H, Amer-Wahlin I, Hagberg H, Herbst A, Kjellmer I, Marsal K, Olofsson P, Rosen KG. Fetal electrocardiography in labor and neonatal outcome: data from the Swedish randomized controlled trial on intrapartum fetal monitoring. Am J Obstet Gynecol. 2003 Jan;188(1):183-92. doi: 10.1067/mob.2003.109. PMID 12548215
- [Background] Neilson JP. Fetal electrocardiogram (ECG) for fetal monitoring during labour. Cochrane Database Syst Rev. 2006 Jul 19;(3):CD000116. doi: 10.1002/14651858.CD000116.pub2. PMID 16855950
- [Background] Amer-Wahlin I, Bordahl P, Eikeland T, Hellsten C, Noren H, Sornes T, Rosen KG. ST analysis of the fetal electrocardiogram during labor: Nordic observational multicenter study. J Matern Fetal Neonatal Med. 2002 Oct;12(4):260-6. doi: 10.1080/jmf.12.4.260.266. PMID 12572595
- [Background] Luttkus AK, Noren H, Stupin JH, Blad S, Arulkumaran S, Erkkola R, Hagberg H, Lenstrup C, Visser GH, Tamazian O, Yli B, Rosen KG, Dudenhausen JW. Fetal scalp pH and ST analysis of the fetal ECG as an adjunct to CTG. A multi-center, observational study. J Perinat Med. 2004;32(6):486-94. doi: 10.1515/JPM.2004.121. PMID 15576269
- [Background] Kwee A, van der Hoorn-van den Beld CW, Veerman J, Dekkers AH, Visser GH. STAN S21 fetal heart monitor for fetal surveillance during labor: an observational study in 637 patients. J Matern Fetal Neonatal Med. 2004 Jun;15(6):400-7. doi: 10.1080/14767050410001727404. PMID 15280112
- [Background] Vayssiere C, Haberstich R, Sebahoun V, David E, Roth E, Langer B. Fetal electrocardiogram ST-segment analysis and prediction of neonatal acidosis. Int J Gynaecol Obstet. 2007 May;97(2):110-4. doi: 10.1016/j.ijgo.2007.01.003. Epub 2007 Mar 26. PMID 17368461
- [Background] Noren H, Blad S, Carlsson A, Flisberg A, Gustavsson A, Lilja H, Wennergren M, Hagberg H. STAN in clinical practice--the outcome of 2 years of regular use in the city of Gothenburg. Am J Obstet Gynecol. 2006 Jul;195(1):7-15. doi: 10.1016/j.ajog.2006.01.108. Epub 2006 Apr 27. PMID 16643829
- [Background] Ross MG, Devoe LD, Rosen KG. ST-segment analysis of the fetal electrocardiogram improves fetal heart rate tracing interpretation and clinical decision making. J Matern Fetal Neonatal Med. 2004 Mar;15(3):181-5. doi: 10.1080/14767050410001668284. PMID 15280144
- [Background] Devoe LD, Ross M, Wilde C, Beal M, Lysikewicz A, Maier J, Vines V, Amer-Wahlin I, Lilja H, Noren H, Maulik D. United States multicenter clinical usage study of the STAN 21 electronic fetal monitoring system. Am J Obstet Gynecol. 2006 Sep;195(3):729-34. doi: 10.1016/j.ajog.2006.06.002. PMID 16949404
- [Background] Macones GA, Hankins GD, Spong CY, Hauth J, Moore T. The 2008 National Institute of Child Health and Human Development workshop report on electronic fetal monitoring: update on definitions, interpretation, and research guidelines. J Obstet Gynecol Neonatal Nurs. 2008 Sep-Oct;37(5):510-5. doi: 10.1111/j.1552-6909.2008.00284.x. PMID 18761565
- [Background] Siggaard-Andersen O. An acid-base chart for arterial blood with normal and pathophysiological reference areas. Scand J Clin Lab Invest. 1971 May;27(3):239-45. doi: 10.3109/00365517109080214. No abstract available. PMID 5581186
- [Background] Shankaran S, Laptook AR, Ehrenkranz RA, Tyson JE, McDonald SA, Donovan EF, Fanaroff AA, Poole WK, Wright LL, Higgins RD, Finer NN, Carlo WA, Duara S, Oh W, Cotten CM, Stevenson DK, Stoll BJ, Lemons JA, Guillet R, Jobe AH; National Institute of Child Health and Human Development Neonatal Research Network. Whole-body hypothermia for neonates with hypoxic-ischemic encephalopathy. N Engl J Med. 2005 Oct 13;353(15):1574-84. doi: 10.1056/NEJMcps050929. PMID 16221780
- [Background] Bloom SL, Spong CY, Thom E, Varner MW, Rouse DJ, Weininger S, Ramin SM, Caritis SN, Peaceman A, Sorokin Y, Sciscione A, Carpenter M, Mercer B, Thorp J, Malone F, Harper M, Iams J, Anderson G; National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Fetal pulse oximetry and cesarean delivery. N Engl J Med. 2006 Nov 23;355(21):2195-202. doi: 10.1056/NEJMoa061170. PMID 17124017
- [Background] Jennison C, Turnbull BW. Statistical approaches to interim monitoring of medical trials: a review and commentary. Statist. Sci. 1990; 229-317.
- [Background] Demets DL. Practical aspects in data monitoring: a brief review. Stat Med. 1987 Oct-Nov;6(7):753-60. doi: 10.1002/sim.4780060706. PMID 3321314
- [Background] Pocock SJ. Group sequential methods in the design and analysis of clinical trials. Biometrika 1977; 64: 191-199.
- [Background] O'Brien PC, Fleming TR. A multiple testing procedure for clinical trials. Biometrics. 1979 Sep;35(3):549-56. PMID 497341
- [Background] Lan KK, DeMets DL. Discrete sequential boundaries for clinical trials. Biometrika 1983; 70: 659-63.
- [Background] Lan KK, Wittes J. The B-value: a tool for monitoring data. Biometrics. 1988 Jun;44(2):579-85. PMID 3390511
- [Background] Pocock SJ. When to stop a clinical trial. BMJ. 1992 Jul 25;305(6847):235-40. doi: 10.1136/bmj.305.6847.235. No abstract available. PMID 1392832
- [Background] Stallones RA. The use and abuse of subgroup analysis in epidemiological research. Prev Med. 1987 Mar;16(2):183-94. doi: 10.1016/0091-7435(87)90082-x. PMID 3295858
- [Background] Yusuf S, Wittes J, Probstfield J, Tyroler HA. Analysis and interpretation of treatment effects in subgroups of patients in randomized clinical trials. JAMA. 1991 Jul 3;266(1):93-8. PMID 2046134
- [Derived] Plunkett BA, Weiner SJ, Saade GR, Belfort MA, Blackwell SC, Thorp JM Jr, Tita ATN, Miller RS, McKenna DS, Chien EKS, Rouse DJ, El-Sayed YY, Sorokin Y, Caritis SN; Eunice Kennedy Shriver National Institute of Child Health Human Development Maternal-Fetal Medicine Units (MFMU) Network*. Maternal Diabetes and Intrapartum Fetal Electrocardiogram. Am J Perinatol. 2024 May;41(S 01):e14-e21. doi: 10.1055/a-1817-5788. Epub 2022 Apr 5. PMID 35381609
- [Derived] Belfort MA, Saade GR, Thom E, Blackwell SC, Reddy UM, Thorp JM Jr, Tita AT, Miller RS, Peaceman AM, McKenna DS, Chien EK, Rouse DJ, Gibbs RS, El-Sayed YY, Sorokin Y, Caritis SN, VanDorsten JP; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. A Randomized Trial of Intrapartum Fetal ECG ST-Segment Analysis. N Engl J Med. 2015 Aug 13;373(7):632-41. doi: 10.1056/NEJMoa1500600. PMID 26267623
- See also: The public website of the NICHD Maternal Fetal Medicine Units (MFMU) Network — http://www.bsc.gwu.edu/mfmu

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Group: S31 monitors in the open mode displayed ECG ST-segment information intended for use when uncertain fetal heart-rate patterns were detected. Management of the labor and delivery for women in this group was dictated by the ST-segment analysis guidelines
- Masked Group: The masked S31 monitors functioned as conventional electronic fetal heart-rate monitors. The care of patients in the masked group was managed at the discretion of the attending physician or midwife.
Period: Overall Study
Arm/Group | Open Group | Masked Group
Started | 5532 | 5576
Completed | 5488 | 5529
Not Completed | 44 | 47
Not completed — Randomization error | 5 | 1
Not completed — Declined to continue participation | 8 | 13
Not completed — Physician Decision | 22 | 24
Not completed — Technical problems | 7 | 6
Not completed — Staff error | 2 | 1
Not completed — Ineligible | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Open Group | Masked Group | Total
Number analyzed (Participants) | 5532 | 5576 | 11108
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.4 (5.9) | 27.2 (5.8) | 27.3 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5532 | 5576 | 11108
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 1326 | 1350 | 2676
  White | 3297 | 3281 | 6578
  Other | 909 | 945 | 1854
Week of pregnancy at randomization [Mean (Standard Deviation); unit: weeks] | 39.4 (1.2) | 39.4 (1.2) | 39.4 (1.2)
Body-mass index before pregnancy [Mean (Standard Deviation); unit: kg/m^2] — Population: Pre-pregnancy BMI was not able to be obtained for all participants.
  kg/m^2
    number analyzed (Participants) | 5498 | 5533 | 11031
    (all) | 27.4 (7.2) | 27.4 (7.0) | 27.4 (7.1)
Educational level [Mean (Standard Deviation); unit: years] — Population: Schooling based on self report. Unable to obtain for all participants.
  years
    number analyzed (Participants) | 5484 | 5516 | 11000
    (all) | 12.8 (2.6) | 12.8 (2.7) | 12.8 (2.6)
Cervical dilation at randomization [Median (Inter-Quartile Range); unit: centimeters] | 5 [4 to 6] | 5 [4 to 6] | 5 [4 to 6]
Type of labor [Count of Participants; unit: Participants]
  Spontaneous | 2259 | 2311 | 4570
  Induced | 3273 | 3265 | 6538
Nulliparous [Count of Participants; unit: Participants] | 2354 | 2373 | 4727

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Primary Composite Outcome
Description: Composite primary outcome of intrapartum fetal death, neonatal death, Apgar score <=3 at 5 minutes, neonatal seizure, umbilical artery blood pH <= 7.05 with base deficit >=12 mmol/L in extra-cellular fluid, intubation for ventilation at delivery, neonatal encelphalopathy
Time Frame: From Delivery through 1 month of age
Population: Umbilical cord artery blood was not able to be obtained from all participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Open Group | Masked Group
Number analyzed (Participants) | 5532 | 5576
Participants | 52 | 40
Statistical Analysis 1: Comparison: Open Group vs Masked Group; Analysis on primary composite outcome as a whole; Test type: Superiority or Other; p = 0.20, Chi-squared; Risk Ratio (RR) = 1.31, 95% CI 2-sided [0.87 to 1.98]

2. Primary Outcome: Number of Intrapartum Fetal Deaths (Primary Outcome Component)
Description: Death of the fetus during the intrapartum period.
Time Frame: During labor and through delivery of the baby
Measure: Count of Participants; unit: Participants
Arm/Group | Open Group | Masked Group
Number analyzed (Participants) | 5532 | 5576
Participants | 0 | 0

3. Primary Outcome: Number of Neonatal Deaths (Primary Outcome Component)
Description: Death of the newborn between delivery and1 month of age
Time Frame: Delivery through1 month of age
Measure: Count of Participants; unit: Participants
Arm/Group | Open Group | Masked Group
Number analyzed (Participants) | 5532 | 5576
Participants | 3 | 1
Statistical Analysis 1: Comparison: Open Group vs Masked Group; Test type: Superiority or Other; p = 0.37, Fisher Exact; Risk Ratio (RR) = 3.02, 95% CI 2-sided [0.31 to 29.1]

4. Primary Outcome: Number of Infants With Apgar Score < = 3 at 5 Minutes (Primary Outcome Component)
Description: The Apgar score is a simple method of quickly assessing the health and vital signs of a newborn baby created by and named after Dr. Virginia Apgar. Apgar testing assesses Appearance, Pulse, Grimace and Activity in a newborn and is typically done at one and five minutes after a baby is born, and it may be repeated at 10, 15, and 20 minutes if the score is low. The five criteria are each scored as 0, 1, or 2 (two being the best), and the total score is calculated by then adding the five values obtained. Agar scores of 0-3 are critically low, 4-6 are below normal, and indicate that the baby likely requires medical intervention, scores of 7+ are considered normal. The lower the Apgar score, the more alert the medical team should be to the possibility of the baby requiring intervention. Some components of the Apgar score are subjective, and there are cases in which a baby requires urgent medical treatment despite having a high Apgar score. The lowest score is 0, the highest score is 10.
Time Frame: 5 minutes after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Open Group | Masked Group
Number analyzed (Participants) | 5532 | 5576
Participants | 17 | 6
Statistical Analysis 1: Comparison: Open Group vs Masked Group; Test type: Superiority or Other; p = 0.02, Chi-squared; Risk Ratio (RR) = 2.86, 95% CI 2-sided [1.13 to 7.24]

5. Primary Outcome: Number of Infants Who Experienced Neonatal Seizure (Primary Outcome Component)
Description: Number of infants who experienced Neonatal Seizure
Time Frame: Birth through hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Open Group | Masked Group
Number analyzed (Participants) | 5532 | 5576
Participants | 3 | 4
Statistical Analysis 1: Comparison: Open Group vs Masked Group; Test type: Superiority or Other; p = 1.0, Fisher Exact; Risk Ratio (RR) = 0.76, 95% CI 2-sided [0.17 to 3.38]

6. Primary Outcome: Number of Infants With Umbilical-artery Blood pH < = 7.05 and Base Deficit in Extracellular Fluid > = 12 mmol/Liter (Primary Outcome Component)
Description: Umbilical-artery blood pH < = 7.05 and base deficit in extracellular fluid > = 12 mmol/liter
Time Frame: Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Open Group | Masked Group
Number analyzed (Participants) | 5362 | 5359
Participants | 3 | 8
Statistical Analysis 1: Comparison: Open Group vs Masked Group; Test type: Superiority or Other; p = 0.13, Chi-squared; Risk Ratio (RR) = 0.37, 95% CI 2-sided [0.10 to 1.41]

7. Primary Outcome: Number of Neonates Intubated for Ventilation at Delivery (Primary Outcome Component)
Description: Neonatal intubation for ventilation in the delivery room
Time Frame: Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Open Group | Masked Group
Number analyzed (Participants) | 5532 | 5576
Participants | 42 | 27
Statistical Analysis 1: Comparison: Open Group vs Masked Group; Test type: Superiority or Other; p = 0.07, Chi-squared; Risk Ratio (RR) = 1.57, 95% CI 2-sided [0.97 to 2.54]

8. Primary Outcome: Number of Infants Experiencing Neonatal Encephalopathy (Primary Outcome Component)
Description: Neonatal encephalopathy experienced between delivery and discharge
Time Frame: Delivery through hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Open Group | Masked Group
Number analyzed (Participants) | 5532 | 5576
Participants | 4 | 5
Statistical Analysis 1: Comparison: Open Group vs Masked Group; Test type: Superiority or Other; p = 1.0, Fisher Exact; Risk Ratio (RR) = 0.81, 95% CI 2-sided [0.22 to 3.00]

9. Secondary Outcome: Number of Participants by Delivery Method
Description: Method of delivery of the baby: spontaneous, vacuum assisted, forceps, cesarean
Time Frame: Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Open Group | Masked Group
Number analyzed (Participants) | 5532 | 5576
Participants
  Spontaneous | 4269 | 4348
  Forceps | 128 | 103
  Vacuum-Assisted | 201 | 224
  Cesarean | 934 | 901
Statistical Analysis 1: Comparison: Open Group vs Masked Group; Test type: Superiority or Other; p = .17, Chi-squared

10. Secondary Outcome: Number of Participants by Indication for Cesarean
Description: indication for the cesarean delivery
Time Frame: At any time from randomization through delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Open Group | Masked Group
Number analyzed (Participants) | 934 | 901
Participants
  Fetal Indication | 287 | 298
  Dystocia | 621 | 583
  Other | 26 | 20
Statistical Analysis 1: Comparison: Open Group vs Masked Group; Test type: Superiority or Other; p = 0.45, Chi-squared — The p value was calculated based on the entire study cohort

11. Secondary Outcome: Number of Participants With an Indication for Forceps or Vacuum Delivery
Description: Indication for delivery by forceps or vacuum
Time Frame: During labor through delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Open Group | Masked Group
Number analyzed (Participants) | 329 | 327
Participants
  Fetal indication | 225 | 218
  Dystocia | 95 | 101
  Other | 9 | 8

12. Secondary Outcome: Median Duration of Labor Post-randomization
Description: Duration of labor in hours after randomization through delivery
Time Frame: Onset of Labor through delivery
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Open Group | Masked Group
Number analyzed (Participants) | 5532 | 5576
Hours | 3.8 [2.1 to 6.4] | 3.9 [2.2 to 6.7]
Statistical Analysis 1: Comparison: Open Group vs Masked Group; Test type: Superiority or Other; p = .32, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Number of Neonates With Shoulder Dystocia During Delivery
Description: Presence of shoulder dystocia during delivery
Time Frame: Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Open Group | Masked Group
Number analyzed (Participants) | 5532 | 5576
Participants | 141 | 158
Statistical Analysis 1: Comparison: Open Group vs Masked Group; Test type: Superiority or Other; p = 0.35, Chi-squared

14. Secondary Outcome: Number of Participants With Chorioamnionitis
Description: Chorioamnionitis
Time Frame: Any time from Randomization through Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Open Group | Masked Group
Number analyzed (Participants) | 5532 | 5576
Participants | 286 | 269
Statistical Analysis 1: Comparison: Open Group vs Masked Group; Test type: Superiority or Other; p = 0.40, Chi-squared

15. Secondary Outcome: Number of Participants Who Had a Postpartum Blood Transfusion
Description: Blood transfusion from delivery and through hospital stay until discharge
Time Frame: Delivery through hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Open Group | Masked Group
Number analyzed (Participants) | 5532 | 5576
Participants | 80 | 74
Statistical Analysis 1: Comparison: Open Group vs Masked Group; Test type: Superiority or Other; p = 0.59, Chi-squared

16. Secondary Outcome: Number of Participants Experiencing Postpartum Endometritis
Description: Postpartum endometritis
Time Frame: Delivery through hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Open Group | Masked Group
Number analyzed (Participants) | 5532 | 5576
Participants | 71 | 88
Statistical Analysis 1: Comparison: Open Group vs Masked Group; Test type: Superiority or Other; p = .19, Chi-squared

17. Secondary Outcome: Median Length of Hospital Stay
Description: Days of stay in the hospital
Time Frame: From admission to labor and delivery through hospital discharge
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Open Group | Masked Group
Number analyzed (Participants) | 5532 | 5576
Days | 2 [2 to 2] | 2 [2 to 2]
Statistical Analysis 1: Comparison: Open Group vs Masked Group; Test type: Superiority or Other; p = 0.77, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: Number of Infants Admitted to Special Care Nursery
Description: Intermediate care nursery or neonatal intensive care (anything more than well-baby nursery)
Time Frame: Delivery and 1 month of age
Measure: Count of Participants; unit: Participants
Arm/Group | Open Group | Masked Group
Number analyzed (Participants) | 5532 | 5576
Participants | 498 | 470
Statistical Analysis 1: Comparison: Open Group vs Masked Group; Test type: Superiority or Other; p = 0.28, Chi-squared

19. Secondary Outcome: Median Apgar Score at 5 Minutes
Description: The Apgar score is a simple method of quickly assessing the health and vital signs of a newborn baby created by and named after Dr. Virginia Apgar. Apgar testing assesses Appearance, Pulse, Grimace and Activity in a newborn and is typically done at one and five minutes after a baby is born, and it may be repeated at 10, 15, and 20 minutes if the score is low. The five criteria are each scored as 0, 1, or 2 (two being the best), and the total score is calculated by then adding the five values obtained. Agar scores of 0-3 are critically low, 4-6 are below normal, and indicate that the baby likely requires medical intervention, scores of 7+ are considered normal. The lower the Apgar score, the more alert the medical team should be to the possibility of the baby requiring intervention. Some components of the Apgar score are subjective, and there are cases in which a baby requires urgent medical treatment despite having a high Apgar score.
Time Frame: 5 minutes after Delivery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Open Group | Masked Group
Number analyzed (Participants) | 5532 | 5576
score on a scale | 9 [9 to 9] | 9 [9 to 9]
Statistical Analysis 1: Comparison: Open Group vs Masked Group; Test type: Superiority or Other; p = 0.54, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Number of Infants With Meconium Aspiration Syndrome
Description: Meconium aspiration syndrome
Time Frame: Delivery through discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Open Group | Masked Group
Number analyzed (Participants) | 5532 | 5576
Participants | 20 | 20
Statistical Analysis 1: Comparison: Open Group vs Masked Group; Test type: Superiority or Other; p = 0.98, Chi-squared

21. Secondary Outcome: Number of Infants With a Major Congenital Malformation
Description: Major congenital malformation
Time Frame: Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Open Group | Masked Group
Number analyzed (Participants) | 5532 | 5576
Participants | 38 | 23
Statistical Analysis 1: Comparison: Open Group vs Masked Group; Test type: Superiority or Other; p = .05, Chi-squared

ADVERSE EVENTS:
Time Frame: Data on adverse events was collected on a continuous basis for each participant from the time of randomization up through the time of hospital discharge.
Arm/Group | Open Group | Masked Group
Serious Adverse Events (participants affected / at risk) | 35/5532 | 21/5576
Other Adverse Events (participants affected / at risk) | 0/5532 | 0/5576
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open Group (N=5532) | Masked Group (N=5576)
Postpartum Hemorrhage (Reproductive system and breast disorders) | 7 | 4
Uterine Rupture (Reproductive system and breast disorders) | 2 | 0
Maternal Infection (bacteremia) (Infections and infestations) | 0 | 1
Maternal Seizure (eclampsia) (Nervous system disorders) | 0 | 1
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Neonatal RDS
Congenital malformation (Congenital, familial and genetic disorders) | 11 | 4
Scalp abscess/pustules (neonatal) (Infections and infestations) | 2 | 2 — From site of fetal ECG clip
Neonatal death (Congenital, familial and genetic disorders) | 3 | 1
Neonatal Encephalopathy (Nervous system disorders) | 1 | 0
Neonatal Seizure (Nervous system disorders) | 2 | 1
Subgaleal hematoma (neonate) (Vascular disorders) | 3 | 3
Brachial plexus injury (Nervous system disorders) | 2 | 1
Infection/sepsis (neonate) (Infections and infestations) | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes